CLINICAL TRIAL: NCT04564976
Title: Can Social Support Figures Enhance Fear Extinction in Patients With Social Anxiety?
Brief Title: Social Support and Reduced Fear Acquisition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Naomi Eisenberger, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SSA
Record Dates: First submitted 2020-09-10; First posted 2020-09-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Fear; Anxiety
Keywords: social support; fear acquisition
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Social Support (Experimental)
  Interventions: Behavioral: Social support image

INTERVENTIONS:
Behavioral: Social support image — An image of a social support figure specific to each participant (provided by the participant) will be present while participants undergo a fear acquisition procedure. Specifically--the image will be presented alongside a neutral image that is either consistently paired with shock (CS+) or never paired with shock (CS-), so that assessment of whether there are differences in fear responding (evaluated via SCR) due the shock pairing can be assessed. This is a typical fear acquisition procedure, and a typical outcome would be for SCR to be higher for the CS+ compared to the CS- toward the end and following the procedure, indicating that the CS+ is now associated with the aversive shock and is bringing about a fear response (in this case indexed by increased sympathetic nervous system activity preparing the body to fight or flee).

SUMMARY:
University of California, Los Angeles researchers will recruit healthy participants and anxious participants (those diagnosed with social anxiety disorder) age 18-55 years old to participate in a study examining whether the ability of social support figure reminders to prevent the acquisition of fear in healthy participants extends to those with anxiety disorders.

After being recruited from the UCLA community (healthy participants, n = 50) or referred by treatment providers at the Anxiety and Depression Research Center at UCLA (anxious participants, n =50) and undergoing a telephone screening and in-person screening, 100 participants will be enrolled in the study. During the experiment, all participants will undergo the same procedures: undergoing fear acquisition procedures--the repeated pairing of a neutral image with a mild electric shock that ultimately leads to the association of threat of shock with the image--in the presence of an image of a social support figure (provided by participants) and an image of a smiling stranger.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 18 and 35
* fluent in English
* no history of mental illness (healthy participants: including anxiety, depression, phobia, or any other mental health related disorder diagnosed by a mental health professional)
* diagnosis of social anxiety disorder (anxious participants: allowed co-morbid disorders include depression, other anxiety disorders, and PTSD)

Exclusion Criteria:

* pregnant or planning to become pregnant during the experiment period
* presence of chronic mental illness (healthy participants: as determined by the report of a past diagnosis of mental illness by a physician or psychologist and/or the prescription of medication related to mental health disorder; including anxiety, depression, phobia, or any other diagnosed psychological disorder)
* presence of non-allowed co-morbid disorders (anxious participants: including, bipolar disorder, psychosis, substance use disorder, neurological disorder, and/or obsessive-compulsive disorder)
* current and regular use of prescription medications related to mental health disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fear response during acquisition indicated by elevated Galvanic Skin Response (GSR) | during acquisition procedure
  presence of fear response as indicated by significantly higher galvanic skin response (GSR: an index of peripheral stress responding) to a previously learned fearful image (CS+) compared to a baseline comparator (CS-: never learned to be fearful).
Fear response post-acquisition indicated by elevated GSR | same session - directly post-acquisition (approximately 5 minutes post procedure)
  presence of fear response as indicated by significantly higher galvanic skin response (GSR: an index of peripheral stress responding) to a previously learned fearful image (CS+) compared to a baseline comparator (CS-: never learned to be fearful).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Department of Psychology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No